CLINICAL TRIAL: NCT04340570
Title: Effect of Medication Management at Home Via Pharmacy Home Televisits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 18-286
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Polypharmacy; Deprescribing; Telemedicine
Keywords: polypharmacy; deprescribing; multiple chronic diseases
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Receives pharmacist home televisit for medication management
  Interventions: Behavioral: Medication management via televisit to home
- Usual Care (No Intervention): Usual care for outpatient medication management

INTERVENTIONS:
Behavioral: Medication management via televisit to home — Pharmacist led home based televisit for medication management
  Arms: Intervention

SUMMARY:
Older Veterans, particularly those with multiple chronic conditions requiring complex medication regimens, are more susceptible to adverse effects of medications. In this study, the investigators will examine the effect of a pharmacist led medication management intervention delivered by home televisit on improving medication use. The investigators anticipate that televisit to home by pharmacist for medication management may enhance use of medications at home by Veterans particularly those with complex medication regimens.

DETAILED DESCRIPTION:
Older adults are more likely to suffer from multiple chronic conditions, to be prescribed multiple medications, and are more susceptible to adverse effects of medications. In addition, older adults often use over-the-counter medications and supplements, further complicating their medication regimen. Complex medication regimens are potentially harmful to older adults due to potential drug interactions, potentially inappropriate prescribing or over-the-counter drug use, and medication non-adherence that may lead to poor control of chronic disease. Interventions aimed at reducing medication discrepancy in the ambulatory clinic setting, such as the review of written medication lists, and implementation of "brown bag" reconciliation (asking patients to bring in all medication bottles for review in the clinic) continues to be challenging and have limited success. Clinical pharmacist led interventions to improve appropriate medication use in older adults, including the application of the START/STOPP criteria, have demonstrated effectiveness in reducing adverse drug events. With the increased capability of VA telemedicine to reach Veteran in their homes, delivering medication management via televisit by clinical pharmacists has the potential to yield similar benefits for a larger number of older Veterans.

Telemedicine is an increasingly vital component within VHA to increase access and improve quality of care. By extending care beyond brick-and-mortar clinics, telemedicine increases the reach of care teams and is more convenient for patients, resulting in improved patient satisfaction. Using the capability of telemedicine to reach patients' homes, the investigators propose to examine the effect of medication management by clinical pharmacists via home video televisits, as home video visits have the potential to provide direct visualization of medications in older adults' homes, thereby reducing medication discrepancy and increasing medication adherence. Pharmacist management for older adult medication regimen may also improve appropriate medication use in older adults through direct pharmacist-patient interview and education. In support of this application, preliminary data from the team of investigators demonstrate acceptability of video televisits by older adults, that there is good uptake by patients and VA providers, and that video televisits into the home are feasible.

In this study, the investigators aim to develop a protocol for pharmacy home televisits for medication management in older adults who have multiple chronic conditions and are on multiple medications. The investigators will then conduct a randomized trial to examine the effect of these televisits on appropriate medication use, medication discrepancies, adherence and adverse drug events. The investigators anticipate that a pharmacist led medication management home televisit intervention will lead to reduction in potentially inappropriate use of medication, reduction in medication discrepancies, increased medication adherence and reduced adverse drug events in older adults compared to older adults receiving usual care. The investigators will also examine the potential challenges in implementing the intervention so that the study findings may inform future implementation.

ELIGIBILITY:
Inclusion Criteria:

* Had at least 1 VA primary care visit within past year
* At least 2 chronic conditions
* At least 5 daily medications

Exclusion Criteria:

* Dementia diagnosis
* Lacks capacity for informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 304 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with Potentially inappropriate medication use | 6 months
  Potentially inappropriate medication use (PIM) assessed by blinded reviewer.

SECONDARY OUTCOMES:
Medication Appropriateness | 6 months
  Measured using Medication Appropriateness Index
Adverse drug events | 6 months
  Assessed from subject survey and chart review and rated as preventable vs. nonpreventable
Medication self efficacy | 6 months
  Measured using patient reported "Medication Understanding Use and Self-Efficacy Scale"

CONTACTS AND LOCATIONS:
Overall Officials: William W Hung, MD AB MPH, Principal Investigator — James J. Peters Veterans Affairs Medical Center; Lauren Rachel Moo, MD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (2):
- United States (2):
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hawley CE, Wagner C, Venegas MD, Genovese N, Triantafylidis LK, McCullough MB, Beizer JL, Hung WW, Moo LR. Connecting the disconnected: Leveraging an in-home team member for video visits for older adults. J Am Geriatr Soc. 2024 May;72(5):1408-1419. doi: 10.1111/jgs.18663. Epub 2023 Nov 13. PMID 37960887
- [Derived] Hossain SR, Samant AN, Balsamo BC, Hawley CE, Zanchelli MC, Zhu C, Venegas MD, Robertson M, McCullough MB, Beizer JL, Boockvar KS, Siu AL, Moo LR, Hung WW. Effect of Medication Management at Home via Pharmacist-Led Home Televisits: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2025 Feb 5;14:e65141. doi: 10.2196/65141. PMID 39908544

DOCUMENTS (1):
  • Informed Consent Form (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT04340570/ICF_000.pdf